CLINICAL TRIAL: NCT02859155
Title: Prognostic Factors Affecting Outcomes in Multivisceral en Bloc Resection for Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: CAIO SERGIO NAHAS (Unknown); SERGIO CARLOS NAHAS (Unknown); Ulysses Ribeiro Junior (Unknown); Carlos Frederico Sparapan Marques (Unknown); Rodrigo Ambar Pinto (Unknown); Antonio Rocco Imperiale (Unknown); Guilherme Cutait Cotti (Unknown); William Carlos Nahas (Unknown); Daher Cezar Chade (Unknown); Dariane Sampaio Piato (Unknown); Fabio Busnardo (Unknown); Ivan Cecconello (Unknown)
Responsible Party: Principal Investigator, Leonardo Alfonso Bustamante, M.D, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07081980
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multiviceral resection colorectal cancer (Other): Multiviceral resection surgery of 2 or more intrabdominal organs en bloc with colorectal cancer
  Interventions: Procedure: Multivisceral en bloc resection surgery

INTERVENTIONS:
Procedure: Multivisceral en bloc resection surgery — Multivisceral en bloc resection for colorectal cancer in advance patients (T4)

SUMMARY:
Determine clinical and pathological factors associated with perioperative morbidity and mortality, and oncological outcomes after multivisceral en bloc resection in patients with colorectal cancer.

DETAILED DESCRIPTION:
Between January/2009 and February/2014, 105 patients with primary colorectal cancer selected for multivisceral resection were selected from a prospective database. Clinical and pathological factors, perioperative morbidity and mortality and outcome were verified from medical records. Estimated local recurrence, and overall survival were compared using the log rank method, and Cox regression analysis was used to determine the independence of the studied parameters.

ELIGIBILITY:
Inclusion Criteria:

* T4 Colorectal cancer -

Exclusion Criteria:

* Non primary Colorectal cancer -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-01; Primary Completion 2014-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Survival | 3 years
  diseases free survival

SECONDARY OUTCOMES:
Recurrence | 3 years
  months after local or systemic recurrence for colorectal cancer

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Nahas CSR, Nahas SC, Ribeiro-Junior U, Bustamante-Lopez L, Marques CFS, Pinto RA, Imperiale AR, Cotti GC, Nahas WC, Chade DC, Piato DS, Busnardo F, Cecconello I. Prognostic factors affecting outcomes in multivisceral en bloc resection for colorectal cancer. Clinics (Sao Paulo). 2017 May;72(5):258-264. doi: 10.6061/clinics/2017(05)01. PMID 28591336